CLINICAL TRIAL: NCT06604624
Title: To Evaluate a Multicenter, Randomized, Open, Positive Parallel Controlled Phase III Clinical Trial of Semaglutide Injection (HD1916) in the Treatment of Obesity
Brief Title: Semaglutide in Treatment of Obesity
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HD1916-003
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Weight Management
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, open, positive parallel controlled phase III clinical trial to compare the efficacy and safety of once-weekly HD1916 and semaglutide injection and to evaluate immunogenicity in obese non-diabetic adults.
Who Masked: Participant
Masking Description: This is a multicenter, randomized, open, positive parallel controlled phase III clinical trial to compare the efficacy and safety of once-weekly HD1916 and semaglutide injection and to evaluate immunogenicity in obese non-diabetic adults.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HD1916 (Experimental): HD1916 will be administered via subcutaneous injection once a week in subjects with obesity.
  Interventions: Drug: HD1916
- semaglutide (Active Comparator): semaglutide will be administered via subcutaneous injection once a week in subjects with obesity.
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: HD1916 — HD1916，0.25mg/0.5mg/1.0mg/1.7mg/2.4mg，SC，once a week
  Arms: HD1916
Drug: semaglutide — semaglutide ，0.25mg/0.5mg/1.0mg/1.7mg/2.4mg，SC，once a week
  Arms: semaglutide

SUMMARY:
This is a multicenter, randomized, open, positive parallel controlled phase III clinical trial to compare the efficacy and safety of once-weekly HD1916 and semaglutide injection and to evaluate immunogenicity in obese non-diabetic adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old (at the time of signing ICF), both male and female;
2. BMI≥28 kg/m^2 during screening;
3. Within 90 days before screening, the weight change range controlled by diet and exercise alone is less than 5% (see section 1.3 for the calculation formula);
4. Voluntarily participate in the trial and sign the informed consent.

Exclusion Criteria:

1. Meet any of the following requirements: (1) HbA1c≥6.5% or fasting venous blood glucose ≥7.0 mmol/L during screening; (2) a history of type 1 or type 2 or a specific type of diabetes;
2. Obesity is caused by drugs or diseases (e.g. Cushing's syndrome, acromegaly, etc.); or weight gain caused by increased non-fat content (e.g. edema);
3. Received (including) drug therapy with GLP-1 receptor agonists (single target, double target, or multiple target) within 90 days prior to screening;
4. Received any other drug or product or treatment within 90 days prior to screening that the investigator determines will affect the assessment of weight efficacy of the trial, including but not limited to drugs or products or treatments that contain overweight/obesity or equivalent meaning in the label indications, hypoglycemic drugs, tricyclic antidepressants, antipsychotic or antiepileptic drugs (such as sodium valproate, citalopram, etc.), systemic use of glucocorticoids, etc.;
5. Previous bariatric metabolic surgery (except for previous liposuction, abdominal plastic surgery, intragastric balloon extraction or duodenal jejunal cannulation extraction > 1 year), or planned to receive any surgical treatment during the trial that might affect the evaluation of weight efficacy;
6. Past allergy or suspected allergy to GLP-1 receptor agonists, or past allergy to investigational drug ingredients;
7. Participated in any other trial and received at least one treatment in the 90 days prior to screening;
8. Thyroid function is unstable or uncontrolled 90 days before screening, or TSH> 6.0 mIU/L or < 0.4 mIU/L at screening;
9. Previous or family history of medullary thyroid carcinoma or multiple endocrine adenomatosis type 2 (MEN-2) before screening;
10. Diagnosis of malignant tumors within 5 years prior to screening (except cured skin basal cell carcinoma or cervical carcinoma in situ);
11. Have any of the following major cardiovascular and cerebrovascular history in the 180 days prior to screening: history of myocardial infarction, coronary angioplasty or bypass surgery, valvular heart disease or heart valve repair, clinically significant and treatment-requiring arrhythmia, unstable angina pectoris, decompensated cardiac insufficiency (NYHA Class III or IV), transient ischemic attack, cerebrovascular accident, etc.;
12. Serious gastrointestinal disease (e.g. abnormal gastric emptying, inflammatory bowel disease) before or during screening;
13. Patients with moderate to severe depression at the time of screening, or the total score of PHQ-9 at the time of screening ≥15 points; or history of other serious mental illness (e.g., schizophrenia, bipolar disorder); or have a history of suicidal thoughts, attempted suicide or suicidal behavior;
14. The presence of any of the following before or during screening: chronic pancreatitis, acute pancreatitis, symptomatic gallbladder disease (except cholecystectomy);
15. Any of the following items should be met during screening: (1) systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg; (2) QTcF interval of ECG >450 ms for male or >470 ms for female; (3) eGFR< 30 mL/min/1.73 m^2, eGFR is calculated according to CKD-EPI formula; (4) ALT or AST > 3× upper limit of normal value; (5) blood amylase or blood lipase > 1.5× the upper limit of normal value; (6) blood triglyceride > 5.7 mmol/L; (7) calcitonin ≥50ng/L (pg/mL); (8) HIV antibody or HCV antibody or HBsAg positive (except for HBsAg positive but HBV DNA quantitative test results are not higher than the upper limit of the test reference range and no anti-HBV drugs are used during screening);
16. A history of drug abuse, drug use or alcohol dependence;
17. Total blood donation ≥400 mL or one-time blood loss ≥400 mL within 90 days before screening;
18. Fertile female subjects are pregnant or lactating at the time of screening, or had positive HCG blood; or fertile male or female subjects and their partners are unable to use effective contraception during the trial period and within 3 months after the end of treatment;
19. Other situations in which the investigator does not consider participation in the study appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Relative percentage change in body weight from baseline at 44 weeks of treatment | Baseline through Week44

SECONDARY OUTCOMES:
Proportion of subjects with a weight loss of ≥5% from baseline at 44 weeks of treatment | Baseline through Week44
Proportion of subjects with a weight loss of ≥10% from baseline at 44 weeks of treatment | Baseline through Week44
Changes in waist circumference from baseline at 44 weeks of treatment | Baseline through Week44
Number of TEAE and SAE cases during the experiment | Week0 through Week44
Changes in pulse from baseline at 44 weeks of treatment | Baseline through Week44
Anti-drug antibodies, neutralizing antibodies (anti-drug antibody positive) | Baseline through Week44

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China